CLINICAL TRIAL: NCT04171674
Title: A Study on Plasma and Pulmonary Pharmacokinetics of High-dose Ceftobiprole Given by Continuous Infusion in Mechanically-ventilated Adult Patients With Severe Community-acquired Pneumonia
Brief Title: Pharmacokinetics of High-dose Ceftobiprole in Community-acquired Pneumonia Under Mechanical Ventilation.
Acronym: PAC CEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Centre Hospitalier Lyon Sud (Other); Hôpital Haut-Lévêque (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIVI/2018/CR-01; 2019-002027-15 (EudraCT Number)
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Pneumonia
Keywords: community-acquired pneumonia
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia | interventions — Therapeutics; ceftobiprole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with high-dose ceftobiprole (Experimental)
  Interventions: Drug: Treatment with high-dose ceftobiprole (500mg loading dose followed by 2.5g under continuos infusion).

INTERVENTIONS:
Drug: Treatment with high-dose ceftobiprole (500mg loading dose followed by 2.5g under continuos infusion). — High-dose ceftobiprole (500mg loading dose) will be administered to patients for 30 minutes followed by 2.5g under continuous infusion for 24 hours.

SUMMARY:
The main aim of the study is to describe plasma pharmacokinetics (PK) and pulmonary diffusion of high-dose ceftobiprole (500 mg loading dose followed by 2.5 g under continuous infusion for 24h) for mechanically-ventilated adult patients with severe community-acquired pneumonia, using population PK modelling.

The secondary aims are :

A- To determine whether the pharmacokinetic / pharmacodynamic (PK/PD) targets can be achieved in the plasma and epithelial lining fluid with the recommended doses of ceftobiprole.

B- To define the optimal dose regimen for ceftobiprole in this population.

C- To evaluate clinical recovery (at Day 3 and Day 8) and microbiological recovery (at Day 3).

D- To evaluate the clinical evolution.

E- To evaluate the clinical and biological tolerance.

DETAILED DESCRIPTION:
Pneumonia is still associated with high morbi-mortality, and rapid treatment with suitable antibiotics is required, i.e. with a broad enough spectrum to cover the activity of all the potentially-incriminated pathogens. These antibiotics must be administered at efficient doses and diffused in sufficient quantity at the infection site.

Unlike other beta-lactams, ceftobiprole is a new-generation broad-spectrum cephalosporin which is active on the majority of pathogens encountered in acute, community-acquired pneumonia (CAP) and also on methicillin-resistant staphylococcus aureus (MRSA) and non-fermenting Gram-negative bacilli (GNB) like pseudomonas aeruginosa. It is indicated for the treatment of CAP and also healthcare-associated pneumonia, other than that acquired under mechanical ventilation.

For any antibiotic administered to critically ill patients it is necessary to ensure that the pharmacokinetic/pharmacodynamic (PK/PD) targets correlated with clinical efficacy can be reached with the recommended doses. The DALI study published in 2014 was the first study to alert on the risk of plasma under-dosing when the standard doses of beta lactams were administered in severely ill patients.

Since then, several PK studies performed in the intensive care unit have confirmed the significant risk of non-optimal doses in this population, linked to physiopathological alterations caused by sepsis. So far there have been no studies specifically aimed at the pharmacokinetics of ceftobiprole in those patients with CAP requiring mechanical ventilation. Furthermore, although there is increasing use in the pharmaceutical industry and in the post-developmental phases of medicines, a population PK analysis to help describe the factors influencing the PK of a molecule and establish new dose regimens optimised for a given population (in this case an ICU population) using Monte Carlo simulations, has never been developed for ceftobiprole given by continuous infusion.

The ultimate aim of so-called adequate antibiotic therapy is to obtain the right therapeutic concentrations at the infection site. During a pulmonary infection, the targeted concentrations of antibiotics in the alveolar liquid must be above the minimal inhibitory concentration value at the end of the dose interval for so-called " time-dependent " antibiotics like cephalosporins. Obtaining these efficient concentrations is often made difficult by the beta-lactams' mediocre pulmonary diffusion and can require an increase in doses in order to reach the PK/PD target at the infection site and/or the use of continuous administration of beta-lactamines. Indeed, this way of administrating is being privileged more and more in order to optimise the time spent above the minimal inhibitory concentration.

This pharmacokinetic study is the first to be carried out among a population of ICU patients and one that focuses on pulmonary diffusion of ceftobiprole for the treatment of severe CAP. The main benefits expected are to determine the most suitable doses of ceftobiprole when this molecule is used to treat ICU patients suffering from CAP. With the help of this population analysis, the main aim of the study is therefore to describe the pharmacokinetics (PK) of the plasma and pulmonary diffusion of ceftobiprole administered at high-dosage (500 mg loading dose followed by 2.5 g under continuous infusion for 24h) for severe community-acquired pneumonia under mechanical ventilation.

The secondary aims are :

A- Determine whether the pharmacokinetic / pharmacodynamic (PK/PD) targets can be achieved in the plasma and epithelial lining fluid with the recommended doses of ceftobiprole.

B- Define the optimal dose regimen for ceftobiprole in this population. C- Evaluate the clinical recovery (at Day 3 and Day 8) and microbiological recovery (at Day 3).

D- Evaluate the clinical evolution. E- Evaluate the clinical and biological tolerance.

ELIGIBILITY:
Inclusion Criteria:

* All patients (or his/her representative for those patients who are unable to express their consent) who have given free, informed consent, and signed the consent form.
* All patients affiliated to or benefitting from a health insurance scheme.
* All patients hospitalised in the intensive care unit with severe acute community-acquired pneumonia requiring the use of mechanical ventilation: this is characterised by signs and symptoms corresponding to an infection of the lower respiratory tract and imaging data corresponding to bacterial pneumonia.The patient has been under mechanical ventilation for less than 24 hours.

Exclusion Criteria:

* Any patient who is already taking part in another interventional study that may influence the main criterion for judgement.
* Any patient who is in the exclusion period determined by another study.
* Any patient under curatorship or guardianship established by a court
* Any patient who is pregnant, about to give birth or breastfeeding.
* Any patient with a contra-indication or allergy to beta-lactams
* Any patient whose survival is estimated at less than 48 hours
* Any patient whose discharge from hospital is planned for 24 hours after admission
* Any patient whose creatinine clearance is estimated at less than 50 ml/min or who is undergoing renal replacement therapy
* Any patient undergoing extracorporeal life support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of ceftobiprole on Day 1 | Day 1
  A blood test is performed upon admission to the Intensive Care Unit, BEFORE beginning antibiotic therapy with Ceftobiprole
Blood test after injection of loading-dose Ceftobiprole (Cmax) for 30 minutes | Day 1 (after the 30-minute injection)
  A 3ml blood sample is taken after injection of 500g of Ceftobiprole for 30 minutes, for pharmacological dosage.
Blood test 2 hours AFTER beginning antibiotic therapy with ceftobiprole | Day 1, 2 hours from start of treatment
  After injection of loading-dose Ceftobiprole (Cmax) for 30 minutes followed by 2.5g by continuous infusion of ceftobiprole, a sample is taken at 2 hours from the start of treatment.
Blood test 6 hours AFTER beginning antibiotic therapy with ceftobiprole | Day 1, 6 hours from start of treatment
  After injection of loading-dose Ceftobiprole (Cmax) for 30 minutes followed by 2.5g by continuous infusion of ceftobiprole, a sample is taken at 6 hours from the start of treatment.
Blood test 8 hours AFTER beginning antibiotic therapy with ceftobiprole | Day 1, 8 hours from start of treatment
  After injection of loading-dose Ceftobiprole (Cmax) for 30 minutes followed by 2.5g by continuous infusion of ceftobiprole, a sample is taken at 8 hours from the start of treatment.
Blood test 12 hours AFTER beginning antibiotic therapy with ceftobiprole | Day 1, 12 hours from start of treatment
  After injection of loading-dose Ceftobiprole (Cmax) for 30 minutes followed by 2.5g by continuous infusion of ceftobiprole, a sample is taken at 12 hours from the start of treatment.
Time 2 blood test on third day of antibiotic therapy with ceftobiprole | Day 3 at Time 2
  Patient is on 2.5g of ceftobiprole by continuous infusion. Samples are taken at regular intervals on Day 3.
Time 6 blood test on third day of antibiotic therapy with ceftobiprole | Day 3 at Time 6
  Patient is on 2.5g of ceftobiprole by continuous infusion. Samples are taken at regular intervals on Day 3.
Time 8 blood test on third day of antibiotic therapy with ceftobiprole | Day 3 at Time 8
  Patient is on 2.5g of ceftobiprole by continuous infusion. Samples are taken at regular intervals on Day 3.
Time 12 blood test on third day of antibiotic therapy with ceftobiprole | Day 3 at Time 12
  Patient is on 2.5g of ceftobiprole by continuous infusion. Samples are taken at regular intervals on Day 3.

SECONDARY OUTCOMES:
Pulmonary concentration of ceftobiprole on Day 3 | On Day 3 of treatment with ceftobiprole
  Pulmonary concentrations of ceftobiprole are measured by bronchoalveolar lavage at the same time as any one of the blood samples are taken on Day 3
Plasma concentration BEFORE treatment | Day 1
  A blood test is performed upon admission to the Intensive Care Unit, BEFORE beginning antibiotic therapy with Ceftobiprole to evaluate plasma concentration.
Plasma concentration AFTER maximum dose of ceftobiprole on Day 1 | Day 1
  Patient has now begun antibiotic therapy with Ceftobiprole and has been injected with 500g of Ceftobiprole for 30 minutes. A blood sample is taken to evaluate plasma concentration.
Plasma concentration after two hours at the steady-state | Day 1
  The dosage of Ceftobiprole has now been reduced. Patient is on 2.5g of ceftobiprole by continuous infusion and plasma concentration is measured after 2 hours.
Plasma concentration after 6 hours at the steady-state | Day 1
  Patient is on 2.5g of ceftobiprole by continuous infusion and plasma concentration is measured after 6 hours.
Plasma concentration after 8 hours at the steady-state | Day 1
  Patient is on 2.5g of ceftobiprole by continuous infusion and plasma concentration is measured after 8 hours.
Plasma concentration after 12 hours at the steady-state | Day 1
  Patient is on 2.5g of ceftobiprole by continuous infusion and plasma concentration is measured after 12 hours.
Plasma concentration at Time 2 on Day 2 of the steady-state | Day 2 at Time 2
  Patient is on 2.5g of ceftobiprole by continuous infusion and plasma concentration is measured at Time 2
Plasma concentration at Time 6 on Day 2 of the steady-state | Day 2 at Time 6
  Patient is on 2.5g of ceftobiprole by continuous infusion and plasma concentration is measured at Time 6
Plasma concentration at Time 8 on Day 2 of the steady-state | Day 2 at Time 8
  Patient is on 2.5g of ceftobiprole by continuous infusion and plasma concentration is measured at Time 8
Plasma concentration at Time 12 on Day 2 of the steady-state | Day 2 at Time 12
  Patient is on 2.5g of ceftobiprole by continuous infusion and plasma concentration is measured at Time 12
Plasma concentration on Day 3 (after end of 24H infusion with ceftobiprole) | Day 3 at Time 2
  3ml blood samples are taken and plasma concentration is measured at regular intervals
Plasma concentration on Day 3 (after end of 24H infusion with ceftobiprole) | Day 3 at Time 6
  3ml blood samples are taken and plasma concentration is measured at regular intervals
Plasma concentration on Day 3 (after end of 24H infusion with ceftobiprole) | Day 3 at Time 8
  3ml blood samples are taken and plasma concentration is measured at regular intervals
Plasma concentration on Day 3 (after end of 24H infusion with ceftobiprole) | Day 3 at Time 12
  3ml blood samples are taken and plasma concentration is measured at regular intervals
Presence or not of Ceftobiprole in the epithelial lining fluid on Day 3 (after end of 24H infusion with ceftobiprole) | Day 3
  A sample of epithelial lining fluid is taken on Day 3 by bronchoalveolar lavage and analyzed.
Dose regimens defined by Monte Carlo simulations | After day 3
  Qualitative, pharmacokinetic modelisation using Pmetrics(r) software
Test of cure on Day 3 | Day 3
  The clinician in charge of the patient evaluates the clinical response as follows :
  Resolution:All signs and symptoms related to infection have disappeared Improvement: Marked or moderate reduction of the seriousness and/or number of signs and symptoms of the infection.
  Failure: Insufficient decrease in signs and symptoms related to the infection. No change in patient's condition. Death, even undetermined.
Test of cure on Day 8 | Day 8
  The clinician in charge of the patient evaluates the clinical response as follows :
  Resolution:All signs and symptoms related to infection have disappeared Improvement: Marked or moderate reduction of the seriousness and/or number of signs and symptoms of the infection.
  Failure: Insufficient decrease in signs and symptoms related to the infection. No change in patient's condition. Death, even undetermined.
Test of microbiological cure on Day 3 | Day 3
  Descriptive and quantitative analysis on a cultivated sample taken via bronchoalveolar lavage on Day 3 to check for presence or not of ceftobiprole in the epithelial lining fluid.
Duration of stay at the intensive care unit. | Day 28
  28 days from the beginning of treatment, the number of days that the patient spent in the ICU are noted in the patient's medical file.
Vital status | Day 28
  28 days from the beginning of treatment, the patient's vital status is noted in the patient's medical file (dead/alive).
Number of days alive without mechanical ventilation | Day 28
  28 days from the beginning of treatment, the number of days that the patient has remained alive without mechanical ventilation is noted from the patient's medical file.
Renal function on Day 1 | Day 1
  Creatinine clearance is measured in ML/min to evaluate the patient's renal function
Renal function on Day 2 | Day 2
  Creatinine clearance is measured in ML/min to evaluate the patient's renal function
Evaluation of renal function on Day 3 | Day 3
  Creatinine clearance is measured in ML/min to evaluate the patient's renal function
Evaluation of renal function on Day 8 | Day 8
  Creatinine clearance is measured in ML/min to evaluate the patient's renal function
Evaluation of liver function on Day 1 | Day 1
  The following measurements are taken in order to evaluate the patient's liver function: albumin level (in g/L) and transaminase doses (ALAT, ASAT).
Evaluation of liver function on Day 2 | Day 2
  The following measurements are taken in order to evaluate the patient's liver function: albumin level (in g/L) and transaminase doses (ALAT, ASAT).
Evaluation of liver function on Day 3 | Day 3
  The following measurements are taken in order to evaluate the patient's liver function: albumin level (in g/L) and transaminase doses (ALAT, ASAT).
Evaluation of liver function on Day 8 | Day 8
  The following measurements are taken in order to evaluate the patient's liver function: albumin level (in g/L) and transaminase doses (ALAT, ASAT).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Lyon Sud,, Pierre-Bénite, Auvergne-Rhône-Alpes
  - CHU de Nîmes, Nîmes, Gard

REFERENCES:
- [Result] Roger C, Allaouchiche B, Quintao De Moraes D, Ulrich Feudjio O, Occean BV, Friggeri A, Lefrant JY, Muller L, Breilh D. Intrapulmonary concentrations of ceftobiprole high doses administered by continuous infusion in critically ill patients with community-acquired pneumonia. J Antimicrob Chemother. 2025 Oct 3;80(10):2644-2653. doi: 10.1093/jac/dkaf267. PMID 40754699